CLINICAL TRIAL: NCT05491122
Title: Investigating the Influence of Fluid Intake on Saliva Cortisol: Diurnal Variation and Acute Response to Psychological Stress in Young Adults
Brief Title: The Influence of Fluid Intake on Daily Biological Rhythm and Mental Performance in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ORION Study 2
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2022-06

CONDITIONS: Healthy; Habitual; Drinking; Stress, Physiological; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be screened to identify habitually low, i.e., total fluid intake: men ≤ 1.6 L/day, women ≤ 1.5 L/day and high i.e., total fluid intake: men ≥ 2.9 L/day, women ≥ 2.5 L/day drinkers. Each subject will undergo two different and consecutive experimental periods: 8 days on habitual fluid intake and a 1-week intervention where the intake of drinking water will either be increased (if habitually low) or decreased (if habitually high). The total fluid intake (TFI) prescriptions during the intervention are derived from the mean TFI of habitually high and habitually low drinkers from a sex, age and country matched population. Specifically, habitually high drinkers will be permitted a TFI of 1.3 L/day and habitually low drinkers will be permitted a TFI of 3.5 L/day for men and 3.3 L/day for women. Participants will be instructed to maintain their usual intake of other beverages i.e., tea/coffee to achieve their target TFI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Habitual period (No Intervention): 8 consecutive days where participants will drink fluids as they do habitually (habitually low TFI = ≤ 1.6 L/day, women ≤ 1.5 L/day, or habitually high TFI = men ≥ 2.9 L/day, women ≥ 2.5 L/day)
- Intervention period (Experimental): 1-week where the fluid intake will be modified. Habitually high drinkers will be permitted a TFI of 1.3 L/day and habitually low drinkers will be permitted a TFI of 3.5 L/day for men and 3.3 L/day for women. Participants will be instructed to maintain their usual intake of other beverages i.e., tea/coffee to achieve their target TFI.
  Interventions: Behavioral: Increasing or decreasing daily total fluid intake

INTERVENTIONS:
Behavioral: Increasing or decreasing daily total fluid intake — 1-week intervention where the intake of drinking water will either be increased (if habitually low) or decreased (if habitually high). The total fluid intake (TFI) prescriptions during the intervention are derived from the mean TFI of habitually high and habitually low drinkers from a sex, age and country matched population. Specifically, habitually high drinkers will be permitted a TFI of 1.3 L/day and habitually low drinkers will be permitted a TFI of 3.5 L/day for men and 3.3 L/day for women. Participants will be instructed to maintain their usual intake of other beverages i.e., tea/coffee to achieve their target TFI. The diurnal saliva cortisol response at rest will be examined at the end of both experimental periods and the saliva cortisol response to an acute psychological stress will be examined at the end of the habitual experimental period only.
  Arms: Intervention period

SUMMARY:
Chronic low water intake may raise the risk of morbidity and mortality by influencing key water regulating hormones (e.g., AVP), which are known to modulate glucoregulation and renal function. For example, AVP stimulates the HPA axis to release the glucocorticoid stress hormone cortisol with potentially far-reaching effects on metabolism, immunity and inflammation. One study observed elevated blood cortisol in a group of low water drinkers, albeit cortisol was measured at one time of day only. However, in the field of psychobiology, researchers have traditionally related more dynamic assessments of cortisol with health outcomes; by evoking cortisol responses to acute standardised laboratory stressors, such as The Trier social stress test. More recently, researchers have appreciated the importance of circadian variability in cortisol levels, by examining influences on, and consequences of individual differences in the diurnal variation of cortisol. The major measurable parameters of the diurnal variation are; the cortisol awakening response (CAR), which is the rise in cortisol during the first 30-45 minutes following awakening, and the diurnal cortisol slope, which is the rate of decline in cortisol levels across the day, from morning to evening. These parameters are considered to reflect different aspects of HPA axis function; with the CAR best reflecting the adrenal capacity to respond to stress and awakening and diurnal slope more indicative of daily cortisol exposure. Although distinct, both blunted CAR and a flattened diurnal cortisol slope appear to be consistent markers of HPA axis dysfunction and related to a variety of poor health outcomes. Therefore, it has been recommended that contemporary research should simultaneously estimate an individual's awakening cortisol responsiveness, and diurnal slope, thereby capturing distinct and important components of HPA axis function. The shared pathways that regulate body water, diurnal variation in cortisol and our response to stress underpin the broad aim of this research programme: to investigate the influence of low and high fluid intake on diurnal cortisol variation and the cortisol response to acute stress.

The aims of this study are to investigate:

1. The influence of a change in water intake behaviour on diurnal saliva cortisol variation as assessed by the CAR (primary outcome)
2. The influence of a change in water intake behaviour on biomarkers of hydration and thirst as assessed by urine osmolality, urine colour and thirst sensation.
3. The influence of habitual low and high total fluid intake on saliva cortisol response to an acute psychological stress (secondary outcome)
4. Investigate the influence of a change in water intake behaviour on plasma biomarkers of hydration as assessed by plasma osmolality and plasma copeptin (exploratory outcome)

ELIGIBILITY:
Inclusion Criteria:

Participants who...

* are free-living, who fully understands and agree to the objectives of the study, who gave signed and dated informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* have read and signed the study informed consent.
* are overtly healthy men and current COC using women (taking COC for at least 3-months and should they be eligible and willing to participate, are happy to continue taking COC during their study participation) aged 18-35 years who engage in <5 hours of physical activity per week (in accordance with previously defined classifications). This information will be obtained during the initial study brief and using the health screening questionnaire.
* have a habitual fluid consumption of ≤ 1.6 L/day OR ≥ 2.9 L/day for men and ≤ 1.5 L/day OR ≥ 2.5 L/day for women, verified by 7-day fluid intake record.
* have a verified UOsm aligned with the following and ≤ 28% day-to-day differences in UOsm; this will be determined during the TFI screening week and familiarisation visit 1: IF habitual low TFI, i.e., TFI ≤ 1.5 L/day for women OR ≤ 1.6 L/day for men have a UOsm ≥ 500 mOsm/kg OR IF habitual high TFI, i.e., TFI ≥ 2.5 L/day for women OR ≥ 2.9 L/day for men have a UOsm < 500 mOsm/kg.
* have access to a domestic fridge at home so that urine samples can be stored prior to laboratory visits.
* have a body mass index (BMI) <30 kg/m2.
* have an IOS or Android smart phone and therefore the ability to download the HidrateSpark and MyFitnessPal mobile applications.

Exclusion Criteria:

Participants who…

* had any surgery or intervention requiring a general anaesthesia in the preceding 4 weeks, or who plans to have one during the study.
* have a history of chronic metabolic or gastrointestinal disease, or gastrointestinal surgery except for appendectomy.
* has chronic or iatrogenic immunodeficiency (e.g., Chemotherapy, HIV).
* present a severe evolutive or chronic pathology (e.g., cancer, tuberculosis, Crohn's disease, cirrhosis, multiple sclerosis, Type I diabetes…).
* have cardiac, respiratory (including asthma) or renal insufficiency, cardiomyopathy, valvopathy and medical history of rheumatic fever.
* are receiving (currently or in the 4 last weeks) systemic treatment or topical treatment likely to interfere with the study parameters; specifically, relating to the stress response (e.g., steroid treatment may influence cortisol response) and hydration regulation (e.g., diuretics). Other excluded medications include antibiotics, intestinal or respiratory antiseptics, anti-rheumatics, antiphlogistics (except aspirin or equivalent at doses preventing from aggregation of platelets or blood clotting), anti-inflammatory and steroids prescribed in chronic inflammatory diseases.
* are taking any treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits (e.g., diuretic, hypolipemic, hypoglycemic treatments).
* have a clinically diagnosed psychiatric disorder.
* have a clinically diagnosed sleeping disorder.
* have a clinically diagnosed gambling addiction.
* are involved in any other clinical study within the preceding month or in the exclusion period after another clinical study.
* changes his/her dietary habits within the preceding 4 weeks (for instance start of a diet high in fibres).
* have a diagnosed eating disorder.
* have a special medicated diet (for obesity, anorexia, metabolic pathology…).
* plan to modify her/his dietary habits.

  •...have a daily total fluid intake of: Men: between 1.6 litres per day and 2.9 litres per day OR Women: between 1.5 litres per day and 2.5 litres per day.
* have a UOsm of (determined during TFI screening week and familiarisation visit 1):Men: <500 mOsm/kg if habitual TFI is ≤ 1.6 L/day or ≥ 500 mOsm/kg if habitual TFI ≥ 2.9 L/day OR Women: <500 mOsm/kg if habitual TFI is ≤ 1.5 L/day or ≥ 500 mOsm/kg if habitual TFI ≥ 2.5 L/day.
* have a day-to-day variation in UOsm >28% (determined during TFI screening week and familiarisation visit 1)
* habitually consume >1.3 L/day of hot beverages i.e., tea, coffee (1.3L equates to 4 average sized mugs) as estimated by a fluid intake record questionnaire.
* consumes ≥ 91 units of alcohol per month (equivalent to more than 3 pints of beer per day or more than 3 large glasses of red wine per day).
* are vulnerable defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (Examples are members of a group with a hierarchical structure linked to the Investigator or to the Sponsor, subordinate laboratory personnel, and employees of the Investigator or of the Sponsor).
* are women not currently on COC i.e., naturally menstruating, or on progestogen only forms of contraception (i.e., IUS, mini-pill, implant, injection).
* are women using COC for <3-months prior to reading the participant information sheet or not planning to continue taking COC during their potential participation in the study.
* are pregnant woman as assessed by a questionnaire or woman planning to become pregnant during the study, breast-feeding woman.
* are expected to be living in the same home as a current participant.
* are a current smoker.
* are not able to answer questionnaires by writing whatever the reason.
* have a loss of personal liberty, by administrative or judicial decision.
* are major but with a legal guardian.
* engage in >5 hours physical activity a week.
* do not have access to a domestic fridge at home so that urine samples can be stored prior to laboratory visits.
* do not have an IOS or Android smart phone and therefore the ability to download the HidrateSpark and MyFitnessPal mobile applications.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Cortisol awakening response (CAR) | Assessed during the first 45 minutes after awakening
  A biomarker for Hypothalamic Pituitary Adrenal activity; a naturally occurring increase in cortisol upon waking, assessed by ELISA

SECONDARY OUTCOMES:
Urine Osmolality | Mid-afternoon urine samples will be collected on days 2, 5, 6 and 7 during the habitual and on days 10, 13 and 14 of the intervention periods. T
  The concentration of osmotic solutes present in the urine, measured using a freezing point depression osmometer;
Change in saliva cortisol to acute psychological stress | Delta changes (increase/ decrease) in cortisol response (calculated by subtracting the baseline cortisol value from the peak post-stress induction level (-30 minutes pre-stress minus 10 minutes post-stress)
  Changes in the concentration of saliva free cortisol assessed by ELISA
Urine colour | Mid-afternoon urine samples will be collected on days 2, 5, 6 and 7 during the habitual and on days 10, 13 and 14 of the intervention periods. T
  urine colour which is a common urinary marker used for assessing hydration status, assessed using a urine colour chart has been developed to assess urine concentration in healthy humans;
Thirst sensation | hirst sensation will be collected for daily for a total of 15 days across the habitual and intervention periods.
  subjective rating of thirst will be obtained from a 0-9 thirst sensation scale (0 = "not thirsty at all" to 9 = "very, very thirsty")

OTHER OUTCOMES:
Wake to bedtime Saliva cortisol slope | Bedtime minus wake-up level divided by total time awake, collected across days 6 & 7 (habitual period) and days 14 & 15 (intervention period
  A biomarker for Hypothalamic Pituitary Adrenal activity; the rate of decline in cortisol concentration across the day, from morning to evening
Heart rate during acute psychological stress | Continuously assessed from 30 minutes before to 60 minutes after the stress tests and control tests]
  Continuous measurement of heart rate will be assessed using a telemetric chest strap.
State anxiety inventory (STAI-S) response to acute psychological stress | Change from baseline (before stress challenge) to after stress challenge (immediately after acute psychological stress and 60 minutes after the test) will be compared.
  assessed using the state scale of the state trait anxiety inventory (STAI-S), consisting of a 20-item scale for measuring the intensity of anxiety as an emotional state (S-Anxiety). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80)
Emotional response to acute psychological stress | Change from baseline (before stress challenge) to after stress challenge (immediately after acute psychological stress and 60 minutes after the test)
  As assessed by the Positive and negative affective schedule (PANAS), this will be used to measure the emotional response to acute psychological stress. The PANAS consists of 10 items for positive affect and 10 items for negative affect, which are answered on a 5-point likert scale (from 1 = "very slightly or not at all all", to 5 = "extremely."). Ratings are summed to a positive and a negative affect score. Separate items for the Positive and negative affect scores range from 10 - 50, higher scores represent higher levels of positive and negative affect separately .
Plasma Osmolality | assessed on day 7 (habitual period) and day 15 (intervention period) will be compared between habitual low and high drinkers and in response to the intervention weeks (increased or decreased water intake)
  A marker of intracellular osmolality, measured using a freezing point depression osmometer
Plasma Copeptin | assessed on day 7 (habitual period) and day 15 (intervention period) will be compared between habitual low and high drinkers and in response to the intervention weeks (increased or decreased water intake)
  the influence of a change in water intake behaviour on plasma copeptin

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Walsh, PHD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No